CLINICAL TRIAL: NCT07346469
Title: Exploring the Effects of Magnesium Ions on Peripheral Neuropathy, Serum Magnesium Ion Concentration,Sleep Quality, and Quality of Life in Patients With Colorectal Cancer Receiving Chemotherapy.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-F(I)-20250330
Record Dates: First submitted 2025-12-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer (CRC); Chemotherapy Induced Peripheral Neuropathy (CIPN); Sleep Quality; Quality of Life (QOL)
Keywords: Colorectal cancer (CRC); Chemotherapy induced peripheral neuropathy (CIPN); Sleep Quality; Quality of life (QOL)
MeSH Terms: conditions — Colorectal Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study employed an experimental design. Experimental group 1 (25 participants) received one packet of oral magnesium ions daily, while experimental group 2 (25 participants) received one packet of oral magnesium ions daily and a foot bath device with magnesium ion solution added for warm water soaking for 10-15 minutes daily. The control group (25 participants) received no interventional measures. The treatment lasted 3-6 months, and changes in blood magnesium ion concentration were measured during routine blood tests at each hospital admission for chemotherapy (data collected a total of 6 times). Research tools included a structured questionnaire: a basic information questionnaire (17 questions), a functional assessment of cancer treatment/gynecologic oncology group - neurotoxicity (FACT/GOG-Ntx) (38 questions), and the Verran and Snyder-Halpern Sleep Scale (VSH) (15 questions), requiring approximately 25 minutes of study time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Comparator (No Intervention): Routine care without interventional measures
- Experimental Group 1 (oral administration of magnesium ions) (Experimental): Take one packet of oral magnesium ions (400mg) daily
  Interventions: Dietary Supplement: oral magnesium ions
- Experimental Group 2 (oral administration of magnesium ions + foot soak in magnesium ion solution) (Experimental): oral magnesium ions (400 mg) daily, and soak your feet in warm water containing soapberry magnesium ions
  Interventions: Combination Product: oral magnesium ions and warm water with Gu Bao Sapindus mukorossi magnesium ion solution

INTERVENTIONS:
Dietary Supplement: oral magnesium ions — Take one packet of oral magnesium ions (400 mg) daily for 3 months until the end of the 6th chemotherapy session.
  Arms: Experimental Group 1 (oral administration of magnesium ions)
Combination Product: oral magnesium ions and warm water with Gu Bao Sapindus mukorossi magnesium ion solution — Take one packet of oral magnesium ions (400 mg) daily, and soak your feet in warm water containing soapberry magnesium ions for 10-15 minutes, continuing for 3 months until the end of the 6th chemotherapy session.
  Arms: Experimental Group 2 (oral administration of magnesium ions + foot soak in magnesium ion solution)

SUMMARY:
Chemotherapy for colorectal cancer (CRC) is frequently complicated by chemotherapy-induced peripheral neuropathy (CIPN) and impaired sleep quality, significantly impacting patient quality of life. Low magnesium levels have been implicated in peripheral nerve dysfunction. This interventional study aims to investigate the effects of magnesium supplementation on serum magnesium concentration, CIPN severity, and sleep quality in CRC patients undergoing chemotherapy.

Study Design and Methods

This is a prospective, parallel-group, randomized controlled trial (RCT) utilizing a longitudinal design. Participants (CRC patients undergoing chemotherapy) will be randomly allocated to one of three groups:

* Experimental Group 1: Oral magnesium (400mg) supplementation.
* Experimental Group 2: Oral magnesium (400mg}) supplementation and magnesium solution foot baths.
* Control Group: Standard care.

Measurements will be collected using structured questionnaires and blood samples during each chemotherapy cycle. The primary outcomes will be assessed using:

* Serum Magnesium Concentration
* CIPN Severity: Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-neurotoxicity (FACT/GOG-Ntx) scale.
* Sleep Quality: Verran and Snyder-Halpern Sleep Scale (VSH). Primary Research Questions (Hypotheses)

  1. Can the magnesium intervention (oral and/or foot baths) effectively increase the serum magnesium concentration in CRC patients?
  2. Can the magnesium intervention alleviate or improve the severity of CIPN?
  3. Can the magnesium intervention improve the sleep quality of CRC patients during chemotherapy? The intervention groups will be compared against the control group to determine if the magnesium interventions lead to superior improvement in the measured outcomes.

DETAILED DESCRIPTION:
(I) Study Main Purpose This study aims to understand the relevant impact and changes of magnesium on peripheral neuropathy during chemotherapy in colorectal cancer patients. Since there is currently no absolutely effective method to prevent the occurrence of peripheral neuropathy, the expected results of this research can provide colorectal cancer patients with an evidence-based method for peripheral neuropathy prevention, thereby improving their quality of life.

(II) Background and Objectives l Overview of Colorectal Cancer (CRC) According to data from the Ministry of Health and Welfare in 2024, malignant tumors have remained the leading cause of death in Taiwan since 1982. Colorectal cancer (CRC) accounts for 13.2% of cancer deaths, ranking second among the top ten major cancer causes. CRC is one of the most common and fatal cancers globally. Its development is often gradual, involving multiple genetic mutations. Based on the adenoma-carcinoma sequence, normal colonic mucosal epithelial cells overproliferate due to the loss of the APC (adenomatous polyposis coli) gene, gradually forming early adenomas. This progresses to CRC due to K-RAS (Kirsten-ras gene) activation and DCC(deleted in colon cancer) gene deletion, subsequently metastasizing to other body parts. The wall of the large intestine consists of the mucosa, submucosa, muscularis propria, subserosa, and serosa. While polyps typically start as benign, prolonged development can lead to a portion becoming cancerous and transforming into CRC. CRC is classified by location: approximately 10% in the cecum, 2% in the ascending colon, 10% in the transverse colon, 3% in the descending colon, 25% in the sigmoid colon, and 50% in the rectum. Over 95% of CRC cases are primarily adenocarcinoma. The incidence of CRC in Taiwan is associated with diet, lifestyle, and heredity, and the incidence in men is approximately 20% to 30% higher than in women.

l Treatment-Related Side Effects and Neuropathy Individuals newly diagnosed with CRC are primarily treated with surgery, often supplemented by radiation therapy and chemotherapy, which may be administered alone or in combination. Side effects of combined chemo- and radiotherapy include oral mucositis, altered taste, dry mouth, nausea, vomiting, fatigue, diarrhea, and peripheral neuropathy, which consequently affect patients' physiological function and quality of life. Chemotherapy has a significant effect on improving the survival rate of CRC. However, patients often suffer long-term side effects from this treatment. Chemotherapy drugs commonly used to treat CRC are highly toxic to the peripheral nervous system. Therefore, patients frequently develop chemotherapy-induced peripheral neuropathy (CIPN). The most common manifestation is sensory neuropathy, leading to severe impairment of dexterity, mobility, and balance. Symptoms include tingling, numbness, and burning pain in the hands or feet, collectively known as Hand-Foot Syndrome (HFS).

The occurrence of HFS causes discomfort in the daily lives of CRC patients, severely impairing their daily activities, including difficulties with fine motor skills, dexterity, mobility, and balance. This impacts patient routines, sleep, and reduces quality of life, potentially leading to dose reduction or even treatment discontinuation. HFS can take six months or more after treatment cessation to slowly improve and disappear, making prevention and continuous management of HFS highly important. Common tools for assessing HFS include the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-neurotoxicity (FACT/GOG-Ntx), the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE), and the Patient Neurotoxicity Questionnaire (PNQ).

l Potential Mechanism of Magnesium in Improving CIPN Neurologist Erick Gamelin proposed that oxalate, a metabolite of oxaliplatin, acts on sodium ion channels or chelates with calcium ions, disrupting the voltage potential and increasing neuronal excitability, leading to nerve damage. Administering calcium and magnesium salt preparations can prevent ion depolarization, thereby preventing neuropathy. Magnesium is crucial for neuromuscular transmission and acts as a membrane stabilizer, influencing both the central and peripheral nervous systems. Its neuroprotective mechanisms include reducing abnormal dorsal root ganglion (DRG) and neuronal degeneration, decreasing oxidative stress, and preventing tissue hypoxia. Therefore, low concentrations of magnesium may be linked to neuropathic pain, especially diabetic neuropathy (DN). Magnesium also acts as an antagonist to the N-methyl-D-aspartate (NMDA) receptor channel, involved in abnormal sensation and pain signal processing. Magnesium is a charged, highly water-soluble ion that cannot directly cross the lipid stratum corneum. It can permeate through essential oils, which loosen the skin barrier, increasing the permeability of water and other molecules, and promoting local blood circulation, indirectly aiding the movement of solutes (like magnesium salts). Studies show that iontophoresis can enhance absorption. A weak direct current in an electric footbath with magnesium solution creates an "electrodriving" effect, pushing magnesium ions towards the skin, increasing the chance for charged particles to be absorbed through the skin in an aqueous medium.

Low magnesium levels are also associated with impaired peripheral nerve function and axonal degeneration, which may exacerbate neuropathy symptoms . Thus, a decrease in magnesium concentration may be a factor leading to the development or worsening of peripheral neuropathy. Furthermore, serum and intracellular magnesium concentrations may be important indicators for predicting the development and future prognosis of peripheral neuropathy; however, current related research is limited, and the correlation between magnesium intervention and improvement in peripheral neuropathy, sleep quality, and quality of life remains insufficiently explored.

(III) Research Gap Colorectal cancer is a common cancer in Taiwan, and while its treatment effectively improves survival, chemotherapy often causes CIPN, leading to symptoms like numbness, tingling, and burning pain in the hands and feet. This subsequently affects daily activities, sleep, and quality of life. Existing studies mainly focus on general discussions of chemotherapy side effects, with limited research on the long-term impact of CIPN and potential methods for improvement.

Recent literature suggests that low magnesium ion concentration is related to nerve function impairment and axonal degeneration, potentially serving as a critical factor in the development or worsening of peripheral neuropathy. However, there is a lack of randomized controlled trials targeting CRC chemotherapy patients to verify whether magnesium supplementation can improve CIPN. Furthermore, although serum and intracellular magnesium concentrations are considered important biomarkers for predicting CIPN development and prognosis, relevant longitudinal follow-up studies are lacking. Crucially, past research has largely focused on symptomatic relief, rarely integrating sleep quality and quality of life into a comprehensive assessment. Therefore, the causal relationship between "Magnesium Intervention - Peripheral Neuropathy - Sleep Quality - Quality of Life" remains unclear.

Based on the aforementioned gaps, this study proposes a randomized controlled trial combined with a longitudinal design to explore the efficacy of magnesium intervention in improving peripheral neuropathy in CRC chemotherapy patients, and further examine changes in serum magnesium concentration, sleep quality, and quality of life. The aim is to provide an important basis for clinical care and patient prognosis assessment.

(IV) Research Methods and Procedure Execution Schedule l Research Design This study adopts a Prospective, Randomized Controlled Trial (RCT) design with a Parallel Group approach, utilizing a Longitudinal Research Design. Data will be collected using structured questionnaires. Subjects enrolled in the study will be assessed by the principal investigator with a questionnaire (T0) and then randomly assigned to Experimental Group 1 (receiving oral magnesium (400mg) once daily), Experimental Group 2 (receiving oral magnesium (400mg) once daily and magnesium solution foot baths), or the Control Group (receiving standard care).

l Execution Site Colorectal Surgery Ward. l Target Population and Sample Size Colorectal cancer patients. The sample size was calculated using G-power 3.1 software with the F test statistical method, selecting the "ANOVA: Repeated measures, within-between interaction" model. Setting a small effect size of 0.3, a Type I error significance level alpha = 0.05, and a statistical power of Power= 0.8, the required effective sample size is 54 individuals (18 per group). Estimating a 20% loss to follow-up within one month, the planned enrollment is 75 participants (25 per group).

l Execution Steps and Methods Inpatients or outpatients diagnosed with CRC who meet the inclusion and exclusion criteria will be approached by the researcher. The researcher will personally explain the study's objectives and procedures to the subjects, ensuring they understand their rights. After consent is obtained, they will sign the informed consent form. This study employs an experimental design. Experimental Group 1 (30 people) will be provided with oral magnesium (400mg) once daily. Experimental Group 2 (30 people) will be provided with oral magnesium (400mg) once daily and will use a foot bath machine with magnesium solution for a warm water foot bath for 10-15 minutes daily. The Control Group (30 people) will receive no interventional measures. The intervention will last 3-6 months. During each hospitalization for chemotherapy, routine blood tests will be conducted, and changes in serum magnesium concentration will be simultaneously examined (Data collection will occur a total of 6 times). Research instruments include a structured questionnaire: Basic Information Survey (17 items), FACT/GOG-Ntx (38 items), and Verran and Snyder-Halpern Sleep Scale (VSH) (15 items), requiring approximately 25 minutes to complete. Questionnaires will be face-to-face interviews conducted by the principal investigator and immediately collected. Patients can fill them out themselves, or the principal investigator can assist in completion after verbal narration.

l Inclusion Criteria (Suitable for participation)

1. Patients pathologically confirmed with a CRC diagnosis.
2. Age > 20 years old.
3. Clear consciousness.
4. Able to communicate without barriers in Mandarin or Taiwanese.
5. Patients receiving or planning to start receiving chemotherapy (Oxaliplatin). l Exclusion Criteria (Cannot participate)

<!-- -->

1. ECOG (Eastern Cooperative Oncology Group) score ≧2.
2. Patients using intravenous nutrition.
3. Patients with pre-existing neuropathy.
4. Presence of skin wounds.
5. Patients with a cardiac pacemaker.
6. Patients with phenylketonuria.
7. Patients with diarrhea.
8. Patients with renal insufficiency.
9. Patients with hypermagnesemia.
10. Patients allergic to the ingredients. l Intervention Protocol For the experimental groups, the intervention will begin at the start of cancer treatment (chemotherapy). The principal investigator or research personnel will initiate the daily regimen: Experimental Group 1 will take oral magnesium (400mg) once daily; Experimental Group 2 will take oral magnesium (400mg) once daily and use a foot bath with magnesium solution for 10-15 minutes daily. The FACT/GOG-Ntx scale and the VSH scale will be used to track changes at the 1st (T1), 4th (T2), 5th (T3), and 6th (T4) treatment cycles, starting from the first treatment cycle.

    l Research Instruments
    1. Basic Information Questionnaire

       This includes two parts:

       • Part 1: Personal Attributes and Health Status:

       o Personal Attributes: Gender, age, educational level, marital status, economic status, employment status, and lifestyle (including diet, bowel habits, and heredity).

       o Health Status: Height, weight, Body Mass Index (BMI), ECOG (Eastern Cooperative Oncology Group) performance status, and other comorbidities.

       • Part 2: Disease Characteristics:

       o Cancer diagnosis name and ICD-10 diagnosis code, tumor staging, date of pathological confirmation, type of cancer treatment, Oxaliplatin dosage, etc.
    2. Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) Scale This instrument, developed in 1998, assesses neurotoxicity (neurotoxicity subscale, Ntx subscale) and general quality of life (FACT-G). The neurotoxicity assessment focuses on layer-specific issues related to activity impairment and neuro-pathic distress (11 items). The entire questionnaire comprises 38 items and is used to measure the degree of neuropathy and its impact on quality of life.

       • Reliability and Validity: Cronbach's alpha is 0.83.
       * Assessment Period: Evaluates the patient's overall condition over the past week (last seven days).
       * Content: Covers aspects related to the patient's cancer treatment function assessment, including physical well-being, social/family well-being, emotional well-being, functional well-being, and the degree of peripheral neuropathy.
       * Scoring: Higher scores on individual items indicate greater severity. The higher the total score, the more severe the symptoms; conversely, a lower total score indicates less obvious symptoms.
    3. Verran and Snyder-Halpern Sleep Scale (VSH) This scale was developed by Snyder-Halpern and Verran (1987).

       • Measurement Method: Uses a 10-centimeter Visual Analogue Scale (VAS) horizontal line.

       • Number of Items: 15 items.

       • Purpose: Assesses the subject's sleep patterns.

       • Reliability and Validity: Cronbach's alpha is 0.82.

       • Content: Each item describes the subject's self-reported perception of sleep quality from the previous night, covering four main categories: sleep segmentation, disturbance, sleep effectiveness, and compensatory sleep.

       • Scoring: Each item ranges from 0 to 100 points. A higher score indicates more severe sleep disturbance, while a lower score indicates better sleep.

       ________________________________________ l Data Analysis and Statistical Methods Data will be organized and filed using Excel, and processed and analyzed using the SPSS 23.0 (Chinese Version) statistical software package.

       Descriptive Statistics
       * Methods: Frequency distribution, percentage, mean, standard deviation (SD), maximum, and minimum values.

       Inferential Statistics

       • Baseline Differences: Independent samples t-tests and Chi-square tests will be used to examine baseline differences in demographic variables across the three groups.
       * Group Comparison and Trend Analysis: Generalized Estimating Equations (GEE) will be utilized to analyze the within-group and between-group trends of change in:
       * Serum magnesium concentration.
       * Hand-Foot Syndrome (Peripheral Neuropathy).
       * Sleep quality.
       * Quality of life.

ELIGIBILITY:
Inclusion Criteria:

* a. Patients diagnosed with colorectal cancer by pathology.
* b. Age ≥ 20 years.
* c. Conscious.
* d. Able to communicate fluently in Mandarin and Taiwanese.
* e. Patients who have received or are expected to begin chemotherapy (Oxaliplatin).

Exclusion Criteria:

* a. ECOG (Eastern Cooperative Oncology Group) ≥2 points.
* b. Patients receiving intravenous nutrition.
* c. Patients with pre-existing neuropathy.
* d. Patients with skin wounds.
* e. Patients with implanted pacemakers.
* f. Patients with phenylketonuria.
* g. Patients with diarrhea.
* h. Patients with renal insufficiency.
* i. Patients with hypermagnesemia.
* j. Patients allergic to any of the ingredients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in magnesium concentration | Measurements were taken at baseline (prior to the first chemotherapy cycle, T0) and subsequently before the start of chemotherapy Cycles 2, 3, 4, 5, and 6; the duration of each cycle was fixed at 14 days.
  Serum magnesium concentrations were monitored throughout the study. A baseline level (T0) was obtained prior to the start of the first chemotherapy cycle, followed by subsequent measurements taken before the start of each cycle from Cycle 2 to Cycle 6 (each cycle lasting 14 days).
Neuropathic symptoms and quality of life assessment | Measurements were taken at baseline (prior to chemotherapy, T0) and subsequently at the end of chemotherapy Cycles 1 (T1), 4 (T2), 5 (T3), and 6 (T4); the duration of each cycle was 14 days.
  The outcome measures of this study consist of two components: neuropathy symptoms and overall quality of life (QoL), both assessed using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) scale.
  1. Neuropathy Symptoms: Evaluated using the Ntx subscale score (ranging from 0 to 44) to assess specific sensory and functional neurotoxicity.
  2. Quality of Life: Measured by the FACT-G total score (ranging from 0 to 108) to assess well-being across physical, social, emotional, and functional domains.
  All assessments will be conducted at five specific timepoints: baseline (pre-chemotherapy, T0), at the end of Cycle 1 (T1), at the end of Cycle 4 (T2), at the end of Cycle 5 (T3), and at the end of Cycle 6 (T4); each chemotherapy cycle is defined as 14 days.
Sleep quality assessment | Measurements were taken at baseline (prior to chemotherapy, T0) and subsequently at the end of chemotherapy Cycles 1 (T1), 4 (T2), 5 (T3), and 6 (T4); the duration of each cycle was 14 days.
  The sleep quality of participants was evaluated using the Verran and Snyder-Halpern (VSH) Sleep Scale. Measured via a Visual Analogue Scale (VAS), the results are reported independently across three dimensions: (1) Sleep Disturbance (assessing sleep onset latency and mid-sleep awakenings), (2) Sleep Effectiveness (assessing sleep quality and depth), and (3) Sleep Supplementation (assessing daytime napping and feelings upon awakening).
  All assessments were conducted at five specific timepoints: baseline (pre-chemotherapy, T0), at the end of Cycle 1 (T1), at the end of Cycle 4 (T2), at the end of Cycle 5 (T3), and at the end of Cycle 6 (T4); each chemotherapy cycle was fixed at a duration of 14 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The research has not yet begun, and subsequent resource sharing has not yet taken this aspect into account. The progress will be determined after the research begins.